CLINICAL TRIAL: NCT01541592
Title: Insulin Resistance and Dietary Fat
Brief Title: Does Class of Dietary Fat Affect Insulin Resistance?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert.H.Nelson, Assistant Professor of Family Medicine and Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 11-000179
Record Dates: First submitted 2012-02-21; First posted 2012-03-01 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Insulin Resistance
Keywords: Insulin resistance; Endothelial dysfunction; saturated fat; monounsaturated fat; polyunsaturated fat
MeSH Terms: conditions — Insulin Resistance | interventions — Dietary Fats

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Saturated fat (Active Comparator): Palm oil (rich in the saturated fat palmitate)
  Interventions: Other: Dietary fat
- Monounsaturated fat (Active Comparator): Olive oil (rich in the monounsaturated fat oleate)
  Interventions: Other: Dietary fat
- Polyunsaturated fat (Active Comparator): Safflower oil (rich in the polyunsaturated fat linoleate)
  Interventions: Other: Dietary fat

INTERVENTIONS:
Other: Dietary fat — On the study day, each participant will receive 100 grams of a randomly assigned fat via a nasoduodenal tube. The oil will be infused at a rate of ~1 tablespoon per hour so that the total infusion time will be 6 hours.

SUMMARY:
It has been shown that intravenous fatty acids given to normal volunteers in the form of heparin and lipid emulsions will cause insulin resistance in a matter of a few hours. It is not known if this same phenomenon can be demonstrated with oral fat. The investigators are specifically interested in whether or not there are differences in the induction of insulin resistance between the 3 main classes of fatty acids (saturated, monounsaturated and polyunsaturated).

The investigators also plan to evaluate endothelial dysfunction and blood pressure; both of which frequently accompany insulin resistance.

DETAILED DESCRIPTION:
Type 2 Diabetes and cardiovascular disease are closely linked. A common abnormality in both conditions is insulin resistance. The primary cause of insulin resistance in not known. A significant question is what dietary components contribute to the development of insulin resistance. Based on epidemiologic data, it seems that the type of dietary fat is a significant contributor to the development of insulin resistance. However, some researchers argue that the main determinant is total amount of fat, not the composition.

This study is intended to determine if the main types of fat (saturated, monounsaturated and polyunsaturated) ingested over a short time can cause insulin resistance in lean, healthy people. It has been demonstrated that 6 hours of intravenous fat infused into lean, healthy subjects can result in insulin resistance, as well as blood pressure elevation and endothelial dysfunction. Whether this is so with oral fat is not known. The question is important because there is debate about whether the type of fat is as important as the quantity of fat in a person's daily diet. Settling this debate will enhance the ability of health care personnel to determine the optimal dietary recommendations.

This study will make use of a high fat diet consisting of vegetable oils high in the 3 main fatty acids in plasma (palmitate, oleate and linoleate). Because large fat loads can cause intestinal discomfort, a feeding tube will be used to bypass the stomach. The 3 oils will be assigned randomly following a base line study with saline 2 weeks prior to the intervention. Our primary endpoint is insulin resistance, which will be measured by a euglycemic, hyperinsulinemic clamp. Secondary measures will include changes in blood pressure and in vascular reactivity as measured by ultrasound after brief occlusion of a forearm vessel. The changes will be compared to baseline and to the other 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Lean,healthy adults 18 - 40
* No chronic medications (birth control pills allowed)
* Weight stable
* Normal fasting labs performed at screening
* Body mass index ≤ 25 kg/M^2 .

Exclusion Criteria:

* Insulin dependent diabetes
* Thyroid disease
* History of diabetes or heart disease
* History of type 2 diabetes in parent or sibling

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Change in Insulin Sensitivity from Baseline at Two Weeks | Average of 2 weeks.
  Insulin sensitivity will be measured twice (once at baseline following a nasoduodenal infusion of saline for 6 hours; two weeks later following a nasoduodenal infusion of a vegetable oil high in one of 3 fatty acids for 6 hours) using a euglycemic, hyperinsulinemic clamp as described by R. DeFronzo. The actual measurement is expressed as a glucose infusion rate.

SECONDARY OUTCOMES:
Change in Endothelial Function from Baseline at Two Weeks | Average of two weeks
  Endothelial function will be measured by measuring the dilation of the brachial artery in the elbow following occlusion by a blood pressure cuff, which is then released. The actual measurement involves use of ultrasound by an investigator experienced with this technique.
Change in Systolic Blood Pressure at Two Weeks | Average of two weeks
  Blood pressure will be measured using a standard automated blood pressure cuff. The measurements will be taken several times during each study day.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Nelson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States